CLINICAL TRIAL: NCT03390101
Title: An International Multicenter, Randomized, Double-blind, Placebo-Controlled Clinical Study of Efficacy and Safety of Two Dosing Regimens of BCD-085 (JSC BIOCAD, Russia) in Patients With Moderate to Severe Plaque Psoriasis
Acronym: BCD-085-7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-085-7
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCD-085 Q2W (Experimental): Patients in this arm (85 subjects) will receive 120 mg BCD-085 (two SC injections, 60 mg in 1.0 mL each). Thus, the drug will be administered on Day 1 of Week 0, Day 1 of Week 1, Day 1 of Week 2 (induction), Day 1 of Week 4, Day 1 of Week 6, Day 1 of Week 8, and Day 1 of Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 1 will be given BCD-085 every 4 weeks through Week 50.
  Interventions: Drug: BCD-085 Q2W
- BCD-085 Q4W (Experimental): Patients in this arm (85 subjects) will receive 120 mg BCD-085 (two SC injections, 60 mg in 1.0 mL each). Thus, the drug will be administered on Day 1 of Week 0, Day 1 of Week 1, Day 1 of Week 2 (induction), Day 1 of Week 6 and Day 1 of Week 10. For the purpose of blind design, patients will receive a placebo (2 injections) on day 1 of week 4 and week 8.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 2 will continue BCD-085 every 4 weeks through Week 50.
  Interventions: Drug: BCD-085 Q4W
- Placebo (Placebo Comparator): Patients in this arm (43 subjects) will be given two SC injections of placebo (1.0 mL each) on Day 1 of Week 0, Day 1 of Week 1, Day 1 of Week 2, Day 1 of Week 4, Day 1 of Week 6, Day 1 of Week 8, and Day 1 of Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 3 will receive BCD-085 on Day 1 of Week 12, Day 1 of Week 13, Day 1 of Week 14 (induction), then every 4 weeks through Week 50.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCD-085 Q2W — In Arm 1, the test drug BCD-085 will be used at a dose of 120 mg given as two SC injections according to the following schedule: once a week for the first 3 weeks (induction treatment) and then once every 2 weeks through Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label patients will receive BCD-085 through week 50. The follow-up will continue through week 54.
  Other Names: BCD-085
  Arms: BCD-085 Q2W
Drug: BCD-085 Q4W — In Arm 2, and then once every 4 weeks through Week 10. On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 2 will be given BCD-085 once every 4 weeks through week 50. The follow-up will continue through week 54.
  Other Names: BCD-085
  Arms: BCD-085 Q4W
Drug: Placebo — In Arm 3, patients will be given two SC injections of placebo (1.0 mL each) according to the following schedule: on Day 1 of weeks 0, 1, 2 and then once every 2 weeks through Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 3 will receive BCD-085 at weeks 12, 13, 14 and then once every 4 weeks through week 50. The follow-up will continue through week 54.
  Arms: Placebo

SUMMARY:
BCD-085 is an innovative drug, a monoclonal antibody against interleukin-17. The toxicity, safety, and pharmacokinetics of BCD-085 were investigated in animals, in phase I clinical study in healthy volunteers, and in phase III clinical study in patients with moderate to severe plaque psoriasis. This clinical study aims at investigating the efficacy and safety of BCD-085 every other week regimen (after induction for the first 3 weeks) versus BCD-085 one per month regimen (after induction for first 3 weeks) versus placebo in patients with moderate to severe plaque psoriasis.

Study purpose:

To investigate the efficacy and safety of BCD-085 versus placebo in patients with moderate to severe plaque psoriasis (psoriasis vulgaris)

Study objectives:

1. To compare the efficacy of BCD-085 every 2 weeks versus BCD-085 every 4 weeks versus placebo, based on the proportion of patients who achieved a PASI75, target sPGA score, and on other secondary efficacy measures.
2. To evaluate the proportion of patients in each study arm who develop adverse events with multiple injections of BCD-085 and placebo. Compare the safety profiles of BCD-085 when used every 4 weeks and when used every 2 weeks.
3. 4. To assess the immunogenicity of BCD-085 defined as the proportion of patients who develop anti-drug antibodies (binding or neutralizing).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give a written and signed informed consent.
2. Men or women at least 18 years old at the time of signing the ICF
3. Moderate to severe plaque psoriasis diagnosed at least 6 months before signing the informed consent form.
4. Patients received at least one course of phototherapy or systemic therapy for psoriasis or are candidates for such treatment according to the investigator.
5. Body surface area (BSA) affected by psoriasis of 10% or greater, the PASI score of 10 or greater, and the sPGA score of 3 or greater at screening.
6. Negative pregnancy urine test in female subjects (no test is required in women who are post-menopausal for at least 2 years and in surgically sterile women).
7. The patient must be able to follow the Protocol procedures (in the investigator's opinion).
8. Patients of childbearing potential and their partners with preserved reproductive function must implement reliable contraceptive methods starting from signing informed consent to 20 weeks after the last dose of the study therapy. This requirement does not apply to the patients after surgical sterilization and to females who are post-menopausal for 2 years or longer. Reliable contraception methods suggest using one barrier method in combination with one of the following: spermicides, intrauterine device/oral contraceptives

Exclusion Criteria:

1. Baseline erythrodermic, pustular, and guttate psoriasis or any other skin diseases (e.g. eczema) that can affect/complicate assessment of psoriasis treatment
2. Use of the following medications:

   * Prior use of monoclonal antibodies targeting IL17 or its receptor
   * Prior use of more than one drug containing monoclonal antibodies or their fragments
   * Prior use of monoclonal antibodies within 12 weeks before signing the informed consent.
   * Any systemic medications for psoriasis (including glucocorticoids, methotrexate, sulfasalazine, cyclosporine, acitretin, mycophenolate mofetil, аpremilast, calcitriol derivatives, etc.) used within 4 weeks before signing the ICF If prior systemic therapy with non-biologics was stopped due to any reasons, the screening period can be extended up to 8 weeks during which no new non-biologics are allowed.
   * Use of phototherapy within 4 weeks before signing the ICF
   * Topical medications for psoriasis used within 2 weeks before signing the ICF
   * Vaccination with live or attenuated vaccines within 8 weeks before signing the ICF
3. Any active systemic infection or recurrent infection at screening/randomization
4. HIV, hepatitis B, hepatitis C, or syphilis
5. Blood biochemistry abnormalities appearing as:

   1. baseline creatinine > 2 × ULN
   2. baseline ALT, AST or alkaline phosphatase > 2.5 × ULN
   3. baseline bilirubin > 1.5 × ULN
6. WBC count < 3.0 × 109/L; ANC < <2.0× 109/L; platelet count < 100 × 109/L, or hemoglobin < 90 g/L at baseline
7. Any psychiatric conditions including severe depressive disorders and/or any history of suicidal thoughts or suicidal attempts ;
8. Signs of clinically significant depression (Beck's score of 16 or more at screening)
9. Alcohol or substance abuse
10. Tuberculosis now or in the past
11. Latent TB infection (positive results of the Diaskintest or QuantiFERON test, or T-spot).
12. Concurrent diseases ongoing at screening that may increase the risk of adverse events during the study or affect the evaluation of psoriasis symptoms (mask, enhance or alter the symptoms of psoriasis, or cause clinical or laboratory signs/symptoms similar to those of psoriasis):

    * active inflammatory diseases or aggravation of chronic inflammatory diseases other than psoriasis
    * Stable angina class III-IV, unstable angina or a history of myocardial infarction within 1 year before signing the informed consent
    * Cardiac failure moderate to severe (NYHA class III-IV)
    * Treatment-resistant hypertension
    * A history of severe asthma or angioedema
    * Moderate to severe respiratory failure, COPD grade ¾
    * Diabetes mellitus with unsatisfactory glycemic control, when the level of glycated hemoglobin HbA1С ≥8% (results are valid if the test was performed at the screening or within 3 months before signing the ICF)
    * The patient has thyrotoxicosis, which persists in the presence of thyreostatic medications, or hypothyroidism despite of the thyroid hormone treatment
    * Systemic autoimmune diseases (including but not limited to SLE, rheumatoid arthritis, ankylosing spondylitis, Crohn's disease, ulcerative colitis, systemic scleroderma, inflammatory myopathy, mixed connective tissue disease , intersection syndrome, etc.)
    * Any other underlying conditions (including but not limited to metabolic, hematologic, hepatic, renal, pulmonary, neurological, endocrine, cardiac, gastrointestinal conditions and infections) that, in the opinion of the investigator, may affect the course of psoriasis, affect the assessment of signs/symptoms of psoriasis, or put patients using the study treatment at additional risk
13. Malignancies with less than 5 years of remission
14. Known severe allergies (anaphylaxis or drug allergy to two or more drug products)
15. Known allergy or intolerance to monoclonal antibody drugs (murine, chimeric, humanized, or human) or any other components of the test drug or comparator
16. Major surgery within 30 days before the screening, or a major surgery being scheduled at any time during the study
17. Severe infections (including those that required hospitalization or parenteral antibacterial/antimycotic/antiprotozoal treatment) within 6 months before signing the ICF
18. Systemic antibacterial/antimycotic/antiprotozoal treatment within 2 months before the signing the ICF
19. More than 4 episodes of respiratory infection within 6 months before signing the ICF
20. Episodes of severe mycoses (histoplasmosis, coccidioidomycosis, blastomycosis, etc.) within 6 months before signing the ICF
21. A history of epileptic attacks or seizures
22. Any concurrent diseases during which, in the investigator's opinion, the study treatment can harm the patient
23. Pregnancy, breastfeeding, or planning for pregnancy while participating in the study
24. Participation in any other clinical study within 3 months before signing the ICF or simultaneous participation in other clinical studies
25. Patients will not be re-enrolled in this study if they were randomized to this study and then discontinue the participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — Vice-president, R&D, International business development BIOCAD
Locations (1):
- BIOCAD, Saint Petersburg, Strelna, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Puig L, Bakulev AL, Kokhan MM, Samtsov AV, Khairutdinov VR, Morozova MA, Zolkin NA, Kuryshev IV, Petrov AN, Artemeva AV, Zinkina-Orikhan AV. Efficacy and Safety of Netakimab, A Novel Anti-IL-17 Monoclonal Antibody, in Patients with Moderate to Severe Plaque Psoriasis. Results of A 54-Week Randomized Double-Blind Placebo-Controlled PLANETA Clinical Trial. Dermatol Ther (Heidelb). 2021 Aug;11(4):1319-1332. doi: 10.1007/s13555-021-00554-4. Epub 2021 May 31. PMID 34060012

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-085 Q2W: Patients in this arm (85 subjects) will receive 120 mg BCD-085 (two SC injections, 60 mg in 1.0 mL each). Thus, the drug will be administered on Day 1 of Week 0, Day 1 of Week 1, Day 1 of Week 2 (induction), Day 1 of Week 4, Day 1 of Week 6, Day 1 of Week 8, and Day 1 of Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 1 will be given BCD-085 every 4 weeks through Week 50.
  BCD-085 Q2W: In Arm 1, the test drug BCD-085 will be used at a dose of 120 mg given as two SC injections according to the following schedule: once a week for the first 3 weeks (induction treatment) and then once every 2 weeks through Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label patients will receive BCD-085 through week 50. The follow-up will continue through week 54.
- BCD-085 Q4W: Patients in this arm (85 subjects) will receive 120 mg BCD-085 (two SC injections, 60 mg in 1.0 mL each). Thus, the drug will be administered on Day 1 of Week 0, Day 1 of Week 1, Day 1 of Week 2 (induction), Day 1 of Week 6 and Day 1 of Week 10. For the purpose of blind design, patients will receive a placebo (2 injections) on day 1 of week 4 and week 8.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 2 will continue BCD-085 every 4 weeks through Week 50.
  BCD-085 Q4W: In Arm 2, and then once every 4 weeks through Week 10. On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 2 will be given BCD-085 once every 4 weeks through week 50. The follow-up will continue through week 54.
- Placebo: Patients in this arm (43 subjects) will be given two SC injections of placebo (1.0 mL each) on Day 1 of Week 0, Day 1 of Week 1, Day 1 of Week 2, Day 1 of Week 4, Day 1 of Week 6, Day 1 of Week 8, and Day 1 of Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 3 will receive BCD-085 on Day 1 of Week 12, Day 1 of Week 13, Day 1 of Week 14 (induction), then every 4 weeks through Week 50.
  Placebo: In Arm 3, patients will be given two SC injections of placebo (1.0 mL each) according to the following schedule: on Day 1 of weeks 0, 1, 2 and then once every 2 weeks through Week 10.
  On Week 12, the treatment efficacy will be assessed with a PASI75 score, and the therapies will be unblinded. During the open-label period, patients from Arm 3 will receive BCD-085 at weeks 12, 13, 14 and then once every 4 weeks through week 50. The follow-up will continue through week 54.
Period: Weeks 0-12
Arm/Group | BCD-085 Q2W | BCD-085 Q4W | Placebo
Started | 85 | 84 | 44
Completed | 85 | 82 | 43
Not Completed | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Weeks 12-54
Arm/Group | BCD-085 Q2W | BCD-085 Q4W | Placebo
Started | 85 | 82 | 43
Completed | 82 | 78 | 41
Not Completed | 3 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-085 Q2W | BCD-085 Q4W | Placebo | Total
Number analyzed (Participants) | 85 | 84 | 44 | 213
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [35 to 49] | 41.5 [32 to 53] | 39 [33 to 53] | 42 [33 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 9 | 57
  Male | 63 | 58 | 35 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 85 | 84 | 44 | 213
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Median (Inter-Quartile Range); unit: kg] | 87.3 [75 to 96.1] | 89.5 [78 to 98] | 83.5 [70 to 95] | 87.3 [75 to 97]
Height [Median (Inter-Quartile Range); unit: cm] | 178 [170 to 184] | 176 [168 to 182] | 175.5 [168 to 180] | 176 [169 to 182]
Body Surface Area Affected by Psoriasis (BSA) [Median (Inter-Quartile Range); unit: percentage of BSA] — The body surface area affected by psoriasis (BSA) is estimated with the palm rule. The area of the human palm without fingers corresponds to about 1% of the body surface.
  percentage of BSA | 20 [13 to 42] | 22 [14.5 to 43] | 22.5 [13 to 44] | 22 [14 to 43]
PASI score [Median (Inter-Quartile Range); unit: score] — The Psoriasis Area and Severity Index (PASI) allows evaluating the extent and severity of skin symptoms of psoriasis. Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI: 0 (no disease) to 72 (maximal disease).
  score | 18.4 [14.2 to 27] | 17.9 [15.1 to 28.6] | 19.7 [16.3 to 29.4] | 18.6 [15 to 28.5]
sPGA score [Median (Inter-Quartile Range); unit: score] — The Static Physician Global Assessment (sPGA) scale is used to assess the psoriatic lesions in a certain patient from 0 (clear) to 5 (very severe). Within each area, the severity is estimated by three criteria (induration, desquamation, and erythema).
  score | 3 [3 to 4] | 4 [3 to 4] | 4 [3 to 4] | 3 [3 to 4]

OUTCOME MEASURES:

1. Primary Outcome: • The Proportion (Number) of Patients in Each Study Arm Who Achieved a PASI 75 at Week 12 of Treatment
Description: The Psoriasis Area and Severity Index (PASI) allows evaluating the extent and severity of skin symptoms of psoriasis. Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI: 0 (no disease) to 72 (maximal disease).
  Relative (percentage) change in PASI score from baseline (screening) is calculated as 100 x (baseline value - time point t value) / (baseline value) PASI 75 indicates a 75% or greater reduction in PASI scores from baseline and is indicative of excellent disease improvement.
Time Frame: week 12
Population: ITT-population (all randomized)
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-085 Q2W | BCD-085 Q4W | Placebo
Number analyzed (Participants) | 85 | 84 | 44
Participants | 66 | 70 | 0

ADVERSE EVENTS:
Time Frame: Weeks 0-12
Description: The safety analysis included the data from all randomized patients.
Arm/Group | BCD-085 Q2W | BCD-085 Q4W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/84 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/85 | 1/84 | 0/44
Other Adverse Events (participants affected / at risk) | 15/85 | 13/84 | 8/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-085 Q2W (N=85) | BCD-085 Q4W (N=84) | Placebo (N=44)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-085 Q2W (N=85) | BCD-085 Q4W (N=84) | Placebo (N=44)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ECG signs of myocardial ischaemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 4 (4) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT03390101/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT03390101/SAP_001.pdf